CLINICAL TRIAL: NCT01679886
Title: Comparison of the Diagnostic Performances of 82Rubidium Positron Emission Tomography and Conventional Scintigraphy With CZT Cameras for Detection of Myocardial Ischemia in a Population of Overweighed Patients and Women
Brief Title: Comparison of Rubidium PET and SPECT With CZT Crystals for Detection of Myocardial Ischemia in Overweighed Patients and Women
Acronym: RUBIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOM 11066
Record Dates: First submitted 2012-09-03; First posted 2012-09-06 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2016-06

CONDITIONS: Myocardial Ischemia
Keywords: Position emission tomography;; Rubidium;; Women;; Overweighted patients
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rubidium PET (Experimental): Rubidium PET
  Interventions: Radiation: Rubidium PET

INTERVENTIONS:
Radiation: Rubidium PET — Rubidium PET

SUMMARY:
The main objective of this study will be to compare the diagnostic performances of 82Rubidium-PET associated to pharmacologic stress (Persantine) to 99mTc-Sestamibi-SPECT with CZT cameras associated to a stress test (exercise, pharmacological, mixed) for detection of myocardial ischemia in a population of overweighed patients on one hand, and women on the other hand, in a population with an intermediate prevalence of coronary artery disease (≥ 3 cardiovascular risk factors in asymptomatic patients or prevalence of CAD ≥ 30 % using the DIAMOND-FORRESTER score in symptomatic patients).

DETAILED DESCRIPTION:
The main objective of this study will be to compare the diagnostic performances of 82Rubidium-PET associated to pharmacologic stress (Persantine) to 99mTc-Sestamibi-SPECT with CZT cameras associated to a stress test (exercise, pharmacological, mixed) for detection of myocardial ischemia in a population of overweighed patients on one hand, and women on the other hand, in a population with an intermediate prevalence of coronary artery disease (≥ 3 cardiovascular risk factors in asymptomatic patients or prevalence of CAD ≥ 30 % using the DIAMOND-FORRESTER score in symptomatic patients).

Secondary objectives. (1) Comparison between the size and intensity of myocardial ischemia quantified using the sum difference score, left ventricular function at stress and at rest, measured with 99mTc-Sestamibi-SPECT with CZT cameras and 82Rubidium-PET.

(2) Comparison between the values of coronary fractional flow reserve measured invasively and noninvasively with 82Rubidium-PET in patients with stenosis ≥ 50 % on coronary angiography.

(3) Comparison of the effective dose caused by radiation exposure with 99mTc-Sestamibi-SPECT with CZT cameras and 82Rubidium-PET.

(4) Comparison of the costs of the two diagnostic strategies in this population of patients.

Inclusion criteria: Overweighed (body mass index ≥ 25) or women addressed in the Department of Nuclear Medicine for diagnostic cardiac scintigraphy with an intermediate pre-test prevalence of CAD (≥ 3 cardiovascular risk factors in asymptomatic patients or prevalence of CAD ≥ 30 % using the DIAMOND-FORRESTER score in symptomatic patients).

Non-inclusion criteria: Pregnant women; contraindication to dipyridamole injection.

Number of patients: 310 patients

Duration of the study. Duration of the study for a patient will be 16 months and 28 months for the first patients. Total duration of the study will be 40 months, including an 24-month inclusion time period.

Primary endpoint: Patients will be classified as positive in case of:

* Myocardial ischemia defined as the presence of coronary stenosis ≥ 50 % on coronary angiography with functional impairment of blood flow confirmed by invasive measurement of coronary flow reserve (fractional flow reserve, FFR < 0.8), or, in absence of measurement of FFR, a critical coronary stenosis confirmed by the validation committee of coronary angiographies.
* In absence of coronary angiography, the presence of cardiovascular event (cardiovascular or unknown cause of death, admission for acute coronary syndrome, unstable angina, myocardial ischemia or coronary revascularization) validated by the endpoint adjudication committee in the year following inclusion of the patient in the study.

Secondary endpoints: (1) Size and intensity of myocardial ischemia quantified using the sum difference score and, left ventricular function at stress and at rest, measured with 99mTc-Sestamibi-SPECT with CZT cameras and 82Rubidium-PET. (2) Values of coronary fractional flow reserve measured invasively and noninvasively with 82Rubidium-PET in patients with stenosis ≥ 50 % on coronary angiography. (3) Effective dose caused by radiation exposure with 99mTc-Sestamibi-SPECT with CZT cameras and 82Rubidium-PET. (4) Costs of the two diagnostic strategies in this population of patients.

ELIGIBILITY:
INCLUSION CRITERIA :

-Overweighed (body mass index ≥ 25) or women addressed in the Department of Nuclear Medicine for diagnostic cardiac scintigraphy with an intermediate pre-test prevalence of CAD (≥ 3 cardiovascular risk factors in asymptomatic patients or prevalence of CAD ≥ 30 % using the DIAMOND-FORRESTER score in symptomatic patients).

EXCLUSION CRITERIA :

* Pregnant women;
* Contraindication to dipyridamole injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2012-09; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Myocardial ischemia | 1 year
  Patients will be classified as positive in case of:
  * Coronary stenosis ≥ 50 % on coronary angiography and fractional flow reserve < 0.8, or, in absence of FFR, a critical coronary stenosis.
  * In absence of coronary angiography, presence of cardiovascular event during the following year.

SECONDARY OUTCOMES:
Size and intensity of myocardial ischemia | 1 year
  1. Size and intensity of myocardial ischemia quantified using the sum difference score,
  2. Left ventricular function at stress and at rest
  3. Values of FFR measured invasively and noninvasively
  4. Effective dose caused by radiation exposure
  5. Costs of the two diagnostic strategies

CONTACTS AND LOCATIONS:
Overall Officials: Dominique LE GULUDEC, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Groupe Hospitalier Bichat - Claude Bernard, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sprauel T, Imbert L, Doyeux K, Perrin M, Claudin M, Roch V, Doyen M, Roth N, Lamash Y, Chequer R, Rouzet F, Hyafil F, Marie PY. Assessment of sestamibi CZT-SPECT reconstructed using deep-learning-based virtual attenuation correction maps according to coronary artery territory and with comparison to rubidium-PET. J Nucl Cardiol. 2025 Jul;49:102226. doi: 10.1016/j.nuclcard.2025.102226. Epub 2025 Apr 19. PMID 40258438
- [Derived] Mimouni M, Bulsei J, Darlington M, Estellat C, Rouzet F, Hyafil F, Durand-Zaleski I; RUBIS Trial Group. Cost-effectiveness of 82-Rubidium PET myocardial perfusion imaging for the diagnosis of myocardial ischemia depending on the prevalence of coronary artery disease. EJNMMI Res. 2023 Feb 8;13(1):9. doi: 10.1186/s13550-023-00954-x. PMID 36752899